CLINICAL TRIAL: NCT03507855
Title: The Effect of a Reduced Noise Environment on the Response Time of the Anesthesia Provider to Auditory and Visual Alarms During Induction and Emergence From General Anesthesia
Brief Title: The Effect of a Reduced Noise Environment on the Response Time of the Anesthesia Provider
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joshua Uffman (Other)
Responsible Party: Sponsor-Investigator, Joshua Uffman, Vice Chair, Department of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB18-00227
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Noise Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noise reduction (Experimental): Reduced operating room personnel, low ambient light and soft background music during induction and emergence from anesthesia.
  Interventions: Other: Reduced noise
- Control (Active Comparator): Normal operating room environment.
  Interventions: Other: Normal

INTERVENTIONS:
Other: Reduced noise — All activity will cease when the patient enters the operating room and nonessential personnel will be removed. Ambient lighting will be reduced and communication devices muted.
  Arms: Noise reduction
Other: Normal — No change in the normal operating room environment.
  Arms: Control

SUMMARY:
This project will investigate whether reduction in ambient light and elimination of noise during induction and emergence from anesthesia influences the response time of the anesthesia provider to auditory and visual alarms when compared to a standard operating room. In addition, the investigators will assess the cumulative level of noise exposure that providers experience during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia providers that have agreed to participate.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Induction response time | Within 5 mins of patient entering the OR
  Response time of the anesthesia provider to the auditory/visual alarm during induction of anesthesia
Emergence response time | Within 5-15 mins after completion of surgery
  Response time of the anesthesia provider to the auditory/visual alarm during emergence from anesthesia

SECONDARY OUTCOMES:
Noise exposure | Average of 30 mins - 3 hrs
  Assess the cumulative level of noise exposure to the anesthesia provider during the entire surgery of a patient

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cartabuke, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Bozych M, Tram NK, Rice-Weimer J, Cartabuke RS, Tobias JD, Huffman J, Mpody C, Uffman JC. Operating Room Noise Environment and Behavior in Children Undergoing General Anesthesia: A Randomized Controlled Trial. Anesthesiol Res Pract. 2024 Aug 16;2024:4838649. doi: 10.1155/2024/4838649. eCollection 2024. PMID 39185368